CLINICAL TRIAL: NCT00603447
Title: Phase 1b Multicenter Dose Escalation Study of Carfilzomib With Lenalidomide and Dexamethasone for Safety and Activity in Relapsed Multiple Myeloma
Brief Title: Phase 1b Multicenter Study of Carfilzomib With Lenalidomide and Dexamethasone in Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PX-171-006
Record Dates: First submitted 2008-01-16; First posted 2008-01-29 (Estimated); Results first posted 2015-06-03 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Relapsed Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carfilzomib + Lenalidomide + Dexamethasone (Experimental): Treatment during Cycles 1 through 12 consisted of carfilzomib (15, 20, or 20/27 mg/m²) on Days 1, 2, 8, 9, 15, and 16; lenalidomide (10, 15, 20, or 25 mg) on Days 1 to 21; and low-dose dexamethasone (40 mg) given 30 minutes to 4 hours before the carfilzomib dose on Days 1, 8, and 15, as well as on Day 22. For Cycles 13 and higher, carfilzomib could be omitted on Days 8 and 9 at the investigator's discretion.
  Interventions: Drug: Carfilzomib; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib for Injection was administered intravenously over 10 minutes on Days 1, 2, 8, 9, 15, and 16 of a 28-day cycle for the first 12 cycles. Each dose of Carfilzomib for Injection was normalized to body surface area.
  Other Names: Kyprolis®
Drug: Lenalidomide — Lenalidomide was administered orally on Days 1 to 21 of each 28-day cycle.
  Other Names: REVLIMID®
Drug: Dexamethasone — Dexamethasone 40 mg orally or intravenous equivalent was administered 30 minutes to 4 hours before carfilzomib on Days 1, 8, and 15, as well as on Day 22 of each 28-day cycle.

SUMMARY:
To evaluate the safety and maximum tolerated dose (MTD) of carfilzomib in combination with lenalidomide and dexamethasone in patients with relapsed multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

Disease related:

1. Symptomatic multiple myeloma
2. Relapsed or progressive disease after at least one but no more than three prior therapeutic treatments or regimens for multiple myeloma
3. Prior therapeutic treatment regimens may have included bortezomib, lenalidomide, and/or thalidomide, among other agents.
4. If previously treated with lenalidomide or bortezomib, the subject must not have progressed during the first 3 months of treatment with the drug and must not have discontinued treatment due to lenalidomide intolerance (bortezomib intolerant subjects may enroll).
5. Measurable disease, as indicated by one or more of the following:

   * Serum M-protein ≥ 0.5 g/dL
   * Urine Bence-Jones protein ≥ 200 mg/24 h
   * If Serum Protein Electrophoresis is felt to be unreliable for routine M-protein measurement (particularly for patients with Immunoglobulin (Ig)A multiple myeloma), then quantitative immunoglobulin levels can be accepted.
6. Prior to enrollment, sites must provide evidence of myeloma progression/relapse, with start and stop dates of the most recent treatment regimen, as well as best tumor response to all prior treatment regimens.

   Demographic
7. Males and females ≥ 18 years of age
8. Life expectancy of more than three months
9. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2

   Laboratory
10. Adequate hepatic function, with bilirubin < 2 times the upper limit of normal (ULN) and alanine aminotransferase (ALT) < 3 times ULN
11. Absolute neutrophil count (ANC) ≥ 1,000/mm³, hemoglobin ≥ 8 gm/dL, platelet count ≥ 50,000/ mm³ (≥ 30 × 10^9/L if myeloma involvement in the bone marrow is > 50%)

    * Screening ANC should be independent of granulocyte- and granulocyte/macrophage colony stimulating factor (G-CSF and GM-CSF) support for at least 1 week and of pegylated G-CSF for at least 2 weeks.
    * Subjects may receive red blood cell (RBC) or platelet transfusions, if clinically indicated, in accordance with institutional guidelines
    * Screening platelet count should be independent of platelet transfusions for at least 2 weeks
12. Calculated or measured creatinine clearance of ≥ 50 mL/minute, calculated using the formula of Cockcroft and Gault [(140 - Age) x Mass (kg) / (72 x creatinine mg/dL)]; multiply result by 0.85 (if female). Other generally accepted calculation methods can be substituted.

    Ethical/Other
13. Written informed consent in accordance with federal, local, and institutional guidelines
14. Females of childbearing potential (FCBP) must agree to ongoing pregnancy testing
15. FCBP* must have a negative serum or urine pregnancy test, with a sensitivity of at least 50 mIU/mL within 10-14 days (US/RevAssist®) or 25 mIU/mL within 7-14 days (Canada/RevAidSM), prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or to use two methods of reliable birth control, including at least one highly effective method AND one additional effective method of birth control (contraception) AT THE SAME TIME, beginning 4 weeks prior to initiating treatment with lenalidomide, during therapy, during therapy delay, and continuing for 4 weeks following discontinuation of lenalidomide therapy. If a hormonal method (birth control pills, injections, patch or implants) or intrauterine device (IUD) is not medically possible for the subject, the subject may use another highly effective method or two barrier methods AT THE SAME TIME.
16. Male subjects must agree to NEVER have unprotected sexual contact with a female who can become pregnant and must agree to either completely abstain from sexual contact with females who are pregnant or are able to become pregnant, or he must use a latex condom EVERY TIME he engages in any sexual contact with females who are pregnant or may become pregnant while he is taking lenalidomide and for 4 weeks after he stops taking the drug, even if he has had a successful vasectomy. The subject must agree to inform his physician if he has had unprotected sexual contact with a female who can become pregnant or if he thinks FOR ANY REASON, that his sexual partner may be pregnant.
17. Male subjects cannot donate semen or sperm while taking lenalidomide.
18. All study participants must be registered into the mandatory RevAssist (US) or RevAid (Canada) programs and be willing and able to comply with the requirements of Rev Assist/RevAid
19. Subjects must adhere to the study visit schedule and other protocol requirements and receive outpatient treatment and laboratory monitoring at the institute that administers the drug
20. Subjects must agree to take enteric-coated aspirin 81-325 mg orally daily, or if history of prior thrombotic disease or allergy to aspirin, must be fully anticoagulated with warfarin (INR 2-3) or be treated with full-dose, low molecular weight heparin, as if to treat deep venous thrombosis (DVT)/pulmonary embolism.

Exclusion Criteria:

Disease related

1. Subjects with non-secretory or hyposecretory multiple myeloma, defined as < 0.5 g/dL M-protein in serum, < 200 mg/24 hr Bence Jones protein in urine, or disease only measured by serum free light chain (FLC)
2. Subjects who never achieved at least a durable minimal response (MR, ≥ 25% reduction in M-protein for at least 6 weeks) on any prior therapy
3. Corticosteroid therapy in a dose equivalent to dexamethasone ≥ 4 mg/day or prednisone ≥ 20 mg/day within 3 weeks prior to first dose
4. Use of any other experimental drug or therapy within 28 days of baseline
5. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
6. Plasma cell leukemia
7. Waldenström's macroglobulinemia
8. Chemotherapy with approved or investigative anticancer therapeutics, including steroid therapy dose as defined above, within 3 weeks prior to first dose
9. Radiation therapy or immunotherapy within 4 weeks prior to first dose; localized radiation therapy within 1 week prior to first dose
10. Planned radiation therapy that occurs after the start of treatment
11. Participation in an investigational therapeutic study within 3 weeks or within 5 drug half-lives (t1/2) prior to first dose, whichever time is greater.

    Concurrent conditions
12. Pregnant or lactating females
13. History of allergy to boron or mannitol
14. Major surgery within 3 weeks prior to first dose
15. Congestive heart failure (New York Heart Association class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention or myocardial infarction in the previous six months
16. Uncontrolled hypertension
17. Acute active infection requiring systemic antibiotics, antivirals, or antifungals within two weeks prior to first dose
18. Known or suspected human immunodeficiency virus (HIV) infection, known HIV seropositivity, or active hepatitis A, B, or C infection
19. Non-hematologic malignancy within the past three years except

    1. adequately treated basal cell or squamous cell skin cancer,
    2. carcinoma in situ of the cervix, or
    3. prostate cancer < Gleason Grade 6 with stable prostate specific antigen (PSA) levels
20. Serious psychiatric or medical conditions that could interfere with treatment
21. Significant neuropathy (Grade 3, Grade 4, or Grade 2 with pain) at the time of the first dose and/or within 14 days before enrollment
22. Contraindication to any of the required concomitant drugs, including proton-pump inhibitor (e.g., lansoprazole), enteric-coated aspirin or other anticoagulant, or if a history of prior thrombotic disease, warfarin or low molecular weight heparin
23. Subjects in whom the required program of oral and intravenous fluid hydration is contraindicated, e.g., due to pre-existing pulmonary, cardiac, or renal impairment
24. Subjects with known or suspected amyloidosis
25. Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis
26. Prior carfilzomib treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2008-05; Primary Completion 2013-05 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (12):
- United States (11):
  - Pacific Shores Medical Group, Long Beach, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cornell University, New York, New York
  - Gabrail Cancer Center, Canton, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutch Cancer Research Center, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Wang M, Martin T, Bensinger W, Alsina M, Siegel DS, Kavalerchik E, Huang M, Orlowski RZ, Niesvizky R. Phase 2 dose-expansion study (PX-171-006) of carfilzomib, lenalidomide, and low-dose dexamethasone in relapsed or progressive multiple myeloma. Blood. 2013 Oct 31;122(18):3122-8. doi: 10.1182/blood-2013-07-511170. Epub 2013 Sep 6. PMID 24014245
- [Derived] Niesvizky R, Martin TG 3rd, Bensinger WI, Alsina M, Siegel DS, Kunkel LA, Wong AF, Lee S, Orlowski RZ, Wang M. Phase Ib dose-escalation study (PX-171-006) of carfilzomib, lenalidomide, and low-dose dexamethasone in relapsed or progressive multiple myeloma. Clin Cancer Res. 2013 Apr 15;19(8):2248-56. doi: 10.1158/1078-0432.CCR-12-3352. Epub 2013 Feb 27. PMID 23447001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label study of carfilzomib (CFZ) given in combination with lenalidomide (LEN) and low-dose dexamethasone (DEX) in patients with relapsed multiple myeloma. The study consisted of a dose-escalation portion and an expansion portion. Participants were treated until disease progression (PD) or unacceptable toxicity.
Pre-assignment Details: In the dose-escalation portion, participants were enrolled in sequential cohorts to determine the maximum tolerated doses (MTD) of carfilzomib and lenalidomide. In the expansion portion either the MTD or the maximum planned dose (MPD) from Cohort 6 (if no MTD was determined) was administered to gain additional safety and efficacy information.
Groups:
- 1: CFZ 15 mg/m² + LEN 10 mg: Treatment during Cycles 1 through 12 consisted of carfilzomib 15 mg/m² on Days 1, 2, 8, 9, 15, and 16; lenalidomide 10 mg on Days 1 to 21; and 40 mg dexamethasone on Days 1, 8, and 15, and 22. For Cycles 13 and higher, carfilzomib could be omitted on Days 8 and 9 at the investigator's discretion.
- 2: CFZ 15 mg/m² + LEN 15 mg: Treatment during Cycles 1 through 12 consisted of carfilzomib 15 mg/m² on Days 1, 2, 8, 9, 15, and 16; lenalidomide 15 mg on Days 1 to 21; and 40 mg dexamethasone on Days 1, 8, and 15, and 22. For Cycles 13 and higher, carfilzomib could be omitted on Days 8 and 9 at the investigator's discretion.
- 3: CFZ 15 mg/m² + LEN 20 mg: Treatment during Cycles 1 through 12 consisted of carfilzomib 15 mg/m² on Days 1, 2, 8, 9, 15, and 16; lenalidomide 20 mg on Days 1 to 21; and 40 mg dexamethasone on Days 1, 8, and 15, and 22. For Cycles 13 and higher, carfilzomib could be omitted on Days 8 and 9 at the investigator's discretion.
- 4: CFZ 20 mg/m² + LEN 20 mg: Treatment during Cycles 1 through 12 consisted of carfilzomib 20 mg/m² on Days 1, 2, 8, 9, 15, and 16; lenalidomide 20 mg on Days 1 to 21; and 40 mg dexamethasone on Days 1, 8, and 15, and 22. For Cycles 13 and higher, carfilzomib could be omitted on Days 8 and 9 at the investigator's discretion.
- 5: CFZ 20 mg/m² + LEN 25 mg: Treatment during Cycles 1 through 12 consisted of carfilzomib 20 mg/m² on Days 1, 2, 8, 9, 15, and 16; lenalidomide 25 mg on Days 1 to 21; and 40 mg dexamethasone on Days 1, 8, and 15 and 22. For Cycles 13 and higher, carfilzomib could be omitted on Days 8 and 9 at the investigator's discretion.
- 6: CFZ 20/27 mg/m² + LEN 25 mg: Treatment consisted of carfilzomib 20 mg/m² on Days 1 and 2 of Cycle 1, followed by 27 mg/m² for the remainder of treatment (Days 8, 9, 15, and 16 of Cycle 1 and Days 1, 2, 8, 9, 15, and 16 for all subsequent cycles); lenalidomide 25 mg on Days 1 to 21; and 40 mg dexamethasone on Days 1, 8, and 15 and 22. For Cycles 13 and higher, carfilzomib could be omitted on Days 8 and 9 at the investigator's discretion.
- 7: CFZ 20/27 mg/m² + LEN 25 mg: In the Expansion portion, treatment consisted of carfilzomib 20 mg/m² on Days 1 and 2 of Cycle 1, followed by 27 mg/m² for the remainder of treatment (Days 8, 9, 15, and 16 of Cycle 1 and Days 1, 2, 8, 9, 15, and 16 for all subsequent cycles); lenalidomide 25 mg on Days 1 to 21; and 40 mg dexamethasone on Days 1, 8, and 15 and 22. For Cycles 13 and higher, carfilzomib could be omitted on Days 8 and 9 at the investigator's discretion.
Period: Overall Study
Arm/Group | 1: CFZ 15 mg/m² + LEN 10 mg | 2: CFZ 15 mg/m² + LEN 15 mg | 3: CFZ 15 mg/m² + LEN 20 mg | 4: CFZ 20 mg/m² + LEN 20 mg | 5: CFZ 20 mg/m² + LEN 25 mg | 6: CFZ 20/27 mg/m² + LEN 25 mg | 7: CFZ 20/27 mg/m² + LEN 25 mg
Started | 6 | 6 | 8 | 6 | 6 | 8 | 44
Completed | 6 (Participants on-going as of 08 May 2013, discontinued due to PD or completed treatment per protocol.) | 3 (Participants on-going as of 08 May 2013, discontinued due to PD or completed treatment per protocol.) | 6 (Participants on-going as of 08 May 2013, discontinued due to PD or completed treatment per protocol.) | 4 (Participants on-going as of 08 May 2013, discontinued due to PD or completed treatment per protocol.) | 1 (Participants on-going as of 08 May 2013, discontinued due to PD or completed treatment per protocol.) | 6 (Participants on-going as of 08 May 2013, discontinued due to PD or completed treatment per protocol.) | 20 (Participants on-going as of 08 May 2013, discontinued due to PD or completed treatment per protocol.)
Not Completed | 0 | 3 | 2 | 2 | 5 | 2 | 24
Not completed — Adverse Event | 0 | 1 | 1 | 2 | 1 | 2 | 10
Not completed — Other | 0 | 0 | 1 | 0 | 3 | 0 | 13
Not completed — Withdrew Consent | 0 | 2 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: CFZ 15 mg/m² + LEN 10 mg | 2: CFZ 15 mg/m² + LEN 15 mg | 3: CFZ 15 mg/m² + LEN 20 mg | 4: CFZ 20 mg/m² + LEN 20 mg | 5: CFZ 20 mg/m² + LEN 25 mg | 6: CFZ 20/27 mg/m² + LEN 25 mg | 7: CFZ 20/27 mg/m² + LEN 25 mg | Total
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 6 | 8 | 44 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (6.65) | 64.2 (12.11) | 55.4 (7.74) | 61.7 (6.68) | 57.7 (9.31) | 65.4 (7.85) | 62.4 (10.75) | 61.9 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 3 | 4 | 3 | 3 | 18 | 36
  Male | 5 | 2 | 5 | 2 | 3 | 5 | 26 | 48
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 0 | 2 | 1 | 2 | 1 | 0 | 3 | 9
  Asian/Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 3
  Caucasian | 6 | 3 | 7 | 2 | 5 | 7 | 34 | 64
  Hispanic | 0 | 0 | 0 | 2 | 0 | 1 | 4 | 7
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a participants disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active; 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, no self-care, confined to bed or chair.
  participants
    0 (Fully active) | 2 | 0 | 3 | 1 | 2 | 2 | 23 | 33
    1 (Restrictive but ambulatory) | 4 | 5 | 5 | 5 | 4 | 6 | 17 | 46
    2 (Ambulatory but unable to work) | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 5
Time Since Diagnosis [Median (Full Range); unit: years] | 3.3 [2 to 4] | 2.4 [2 to 5] | 3.9 [2 to 15] | 2.8 [0 to 9] | 3.5 [1 to 22] | 4.3 [1 to 12] | 2.8 [0 to 16] | 3.1 [0 to 22]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Treatment-related are those AEs with possible or probable relationship to carfilzomib, lenalidomide or dexamethasone as assessed by the Investigator. The severity of each adverse event was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 3.0, per the following: Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening and Grade 5 = Death.
  Serious adverse events were defined as AEs meeting one of the following: death, life-threatening, required or prolonged in-patient hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect in the offspring of an exposed participant, important medical events that may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed above, or pregnancy or suspected pregnancy.
Time Frame: From the first dose of study drug until 30 days after the last dose; 1 to 52 months, with an average of 12 months.
Population: Safety population consisting of all treated participants
Measure: Number; unit: participants
Arm/Group | 1: CFZ 15 mg/m² + LEN 10 mg | 2: CFZ 15 mg/m² + LEN 15 mg | 3: CFZ 15 mg/m² + LEN 20 mg | 4: CFZ 20 mg/m² + LEN 20 mg | 5: CFZ 20 mg/m² + LEN 25 mg | 6: CFZ 20/27 mg/m² + LEN 25 mg | 7: CFZ 20/27 mg/m² + LEN 25 mg
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 6 | 8 | 44
participants
  Any adverse event | 6 | 6 | 8 | 6 | 6 | 8 | 44
  Treatment-related adverse event | 4 | 5 | 8 | 4 | 6 | 8 | 43
  Grade 3 or higher adverse event | 5 | 6 | 8 | 6 | 6 | 8 | 41
  Treatment-related Grade 3 or higher adverse event | 1 | 4 | 7 | 4 | 6 | 8 | 38
  Serious adverse event | 3 | 3 | 4 | 4 | 3 | 6 | 22
  AE leading to discontinuation of any study drug | 1 | 1 | 3 | 4 | 2 | 3 | 18
  AE leading to discontinuation of carfilzomib | 0 | 0 | 1 | 2 | 1 | 1 | 9
  Deaths within 30 days of last dose of study drug | 0 | 0 | 0 | 0 | 0 | 0 | 3

2. Primary Outcome: Number of Participants With Dose-limiting Toxicities
Description: Dose-limiting toxicity was defined as any of the following events assessed as related to carfilzomib, lenalidomide, or dexamethasone: Nonhematologic
  * ≥ Grade 2 neuropathy with pain
  * ≥ Grade 3 nonhematologic toxicity (excluding nausea, vomiting, diarrhea, hyperglycemia due to dexamethasone, and rash due to lenalidomide)
  * ≥ Grade 3 nausea, vomiting, or diarrhea uncontrolled by maximal supportive therapy
  * ≥ Grade 4 fatigue persisting > 7 days
  * Treatment delay for toxicity > 21 days
  Hematologic
  * Grade 4 neutropenia (absolute neutrophil count [ANC] < 500/mm³) > 7 days
  * Febrile neutropenia (ANC < 1,000/mm³ with fever ≥ 38.3ºC)
  * Grade 4 thrombocytopenia (platelets < 25,000/mm³) for > 7 days despite holding treatment, or Grade 3 or 4 thrombocytopenia associated with bleeding
  * Treatment delay for toxicity > 21 days.
  The maximum-tolerated dose was defined as the dose level below which a drug-related DLT was observed in ≥ 33% of participants in a cohort.
Time Frame: Cycle 1, 28 days
Population: Safety population for the dose escalation portion of the study
Measure: Number; unit: participants
Arm/Group | 1: CFZ 15 mg/m² + LEN 10 mg | 2: CFZ 15 mg/m² + LEN 15 mg | 3: CFZ 15 mg/m² + LEN 20 mg | 4: CFZ 20 mg/m² + LEN 20 mg | 5: CFZ 20 mg/m² + LEN 25 mg | 6: CFZ 20/27 mg/m² + LEN 25 mg
Number analyzed (Participants) | 6 | 6 | 8 | 6 | 6 | 8
participants | 0 | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: From the first dose of study drug until 30 days after the last dose; 1 to 52 months, with an average of 12 months.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | 1: CFZ 15 mg/m² + LEN 10 mg | 2: CFZ 15 mg/m² + LEN 15 mg | 3: CFZ 15 mg/m² + LEN 20 mg | 4: CFZ 20 mg/m² + LEN 20 mg | 5: CFZ 20 mg/m² + LEN 25 mg | 6: CFZ 20/27 mg/m² + LEN 25 mg | 7: CFZ 20/27 mg/m² + LEN 25 mg
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 4/8 | 4/6 | 3/6 | 6/8 | 22/44
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 8/8 | 6/6 | 6/6 | 8/8 | 42/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1: CFZ 15 mg/m² + LEN 10 mg (N=6) | 2: CFZ 15 mg/m² + LEN 15 mg (N=6) | 3: CFZ 15 mg/m² + LEN 20 mg (N=8) | 4: CFZ 20 mg/m² + LEN 20 mg (N=6) | 5: CFZ 20 mg/m² + LEN 25 mg (N=6) | 6: CFZ 20/27 mg/m² + LEN 25 mg (N=8) | 7: CFZ 20/27 mg/m² + LEN 25 mg (N=44)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colonic stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1
Abscess jaw (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 2 | 3
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngeal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1: CFZ 15 mg/m² + LEN 10 mg (N=6) | 2: CFZ 15 mg/m² + LEN 15 mg (N=6) | 3: CFZ 15 mg/m² + LEN 20 mg (N=8) | 4: CFZ 20 mg/m² + LEN 20 mg (N=6) | 5: CFZ 20 mg/m² + LEN 25 mg (N=6) | 6: CFZ 20/27 mg/m² + LEN 25 mg (N=8) | 7: CFZ 20/27 mg/m² + LEN 25 mg (N=44)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 6 | 2 | 3 | 3 | 14
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 1 | 1 | 1 | 2 | 9
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 3 | 2 | 1 | 0 | 5 | 22
Neutropenia (Blood and lymphatic system disorders) | 4 | 4 | 4 | 2 | 5 | 3 | 16
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3 | 2 | 2 | 3 | 3 | 13
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 4
Ventricular hypertrophy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Corneal lesion (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 2
Eye haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye pain (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 1 | 3 | 1 | 1 | 1 | 6
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 1 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 2 | 2 | 1 | 3 | 11
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 3 | 3 | 4 | 4 | 26
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Gingival swelling (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 1 | 2 | 1 | 2 | 16
Oesophageal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Oral soft tissue disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Palatal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 4
Vomiting (Gastrointestinal disorders) | 0 | 2 | 2 | 2 | 0 | 1 | 11
Asthenia (General disorders) | 2 | 0 | 3 | 0 | 1 | 2 | 5
Axillary pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Catheter site haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Chills (General disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 5
Cyst (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1
Face oedema (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 4 | 5 | 3 | 4 | 6 | 30
Feeling hot and cold (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeling jittery (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Feeling of body temperature change (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2
Influenza like illness (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2
Infusion site bruising (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Injection site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Injection site irritation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 4
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 4 | 2 | 0 | 3 | 2 | 17
Pain (General disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 4
Pitting oedema (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 3
Pyrexia (General disorders) | 0 | 1 | 5 | 3 | 1 | 4 | 19
Temperature intolerance (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haemorrhage (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 3
Eye infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1 | 1 | 0 | 0 | 8
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 4
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 4 | 0 | 0 | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 4 | 1 | 0 | 4 | 19
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 3
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 2 | 0 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Incision site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 7
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 6
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 3
Blood calcium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 4
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 3
Heart rate irregular (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 2 | 0 | 3
Weight increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 1 | 0 | 7
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 1 | 1 | 0 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 5
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 3 | 2 | 3 | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 2
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 2 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3 | 3 | 2 | 1 | 1 | 12
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 1 | 2 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 1 | 1 | 3 | 5
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 0 | 1 | 4 | 16
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 1 | 0 | 1 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 3 | 1 | 2 | 1 | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 6
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 4 | 4 | 1 | 1 | 3 | 17
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 4 | 1 | 1 | 2 | 11
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 4
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 3 | 1 | 2 | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Areflexia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 2 | 1 | 2 | 1 | 6
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 5
Dysstasia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 3 | 2 | 0 | 11
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 2 | 1 | 0 | 1 | 8
Hyporeflexia (Nervous system disorders) | 2 | 2 | 1 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 1
Nerve compression (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuropathic pain (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 5
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 12
Paraesthesia (Nervous system disorders) | 2 | 3 | 2 | 0 | 0 | 3 | 9
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 4
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 4
Affect lability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 3
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 7
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 4
Insomnia (Psychiatric disorders) | 1 | 3 | 3 | 0 | 1 | 1 | 17
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Mood swings (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 2
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5 | 3 | 2 | 3 | 4 | 17
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 3 | 2 | 3 | 3 | 15
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 7
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 12
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 7
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 6
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0 | 1 | 0 | 11
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 3
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 4
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 5
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 4 | 1 | 2 | 2 | 8
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Skin fragility (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 5
Flushing (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 4
Peripheral coldness (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Post thrombotic syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2
Vascular fragility (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.